CLINICAL TRIAL: NCT01833455
Title: The Effects of PVC Suppression on Blood Pressure Control in Patients With Frequent PVCs
Brief Title: Premature Ventricular Contractions (PVCs) and Blood Pressure Control
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment.
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UW-PVC-2012-0510
Record Dates: First submitted 2013-04-09; First posted 2013-04-16 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-01

CONDITIONS: Ventricular Premature Complexes; Blood Pressure
MeSH Terms: conditions — Ventricular Premature Complexes | interventions — Flecainide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PVC Suppression then Placebo (Placebo Comparator): This arm will undergo attempted PVC suppression using flecainide for 28 days and then undergo no PVC suppression using placebo for 28 days.
  Interventions: Drug: PVC Suppression using Flecainide; Drug: No PVC Suppression using Placebo
- Placebo then PVC Suppression (Placebo Comparator): This arm will undergo no PVC suppression using placebo for 28 days and then undergo attempted PVC suppression using flecainide for 28 days.
  Interventions: Drug: PVC Suppression using Flecainide; Drug: No PVC Suppression using Placebo

INTERVENTIONS:
Drug: PVC Suppression using Flecainide — Flecainide will be administered to result in a reduction in PVC burden.
  Other Names: Tambocor
Drug: No PVC Suppression using Placebo — Placebo (sugar pills) will be given to result in no alteration in PVC burden.

SUMMARY:
The purpose of this study is to determine if reduction in premature ventricular contraction (PVC) burden results in a decrease in blood pressure, sympathetic outflow, plasma catecholamines and an improvement in baroreflex gain. Flecainide will be used for PVC suppression in a randomized, double-blinded, crossover fashion.

ELIGIBILITY:
Inclusion Criteria:

* Frequent symptomatic premature ventricular contractions (PVCs) (>10% of total QRSs on a 24-hour Holter)
* Willingness to participate in research

Exclusion Criteria:

* Age > 65 years old
* Pacemaker implantation
* Implantable cardioverter defibrillator implantation requiring pacing
* Sick sinus syndrome
* Atrio-ventricular (AV) block
* Left ventricular dysfunction defined as left ventricular ejection fraction < 50%
* History of myocardial infarction or coronary artery disease
* Severe left ventricular hypertrophy (wall thickness > 1.5 cm by echocardiography performed within 3 months from enrollment)
* Severe liver dysfunction
* Creatinine clearance of 35 mL/min/1.73 square meters or less
* Pregnancy
* Known hypersensitivity to the drug
* QRS duration > 120 ms
* Recent change in blood pressure medication within 30 days of enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Hamdan, MD, MBA, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PVC Suppression Then Placebo | Placebo Then PVC Suppression
Started | 4 | 4
Completed 1st Baseline | 4 | 4
Completed 1st Intervention | 3 | 4
Completed 2nd Baseline (Washout) | 3 | 4
Completed | 3 | 4
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PVC Suppression Then Placebo | Placebo Then PVC Suppression | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 0 | 4
  Male | 0 | 4 | 4
PVC Burden [Mean (Standard Deviation); unit: % of heartbeats] | 26 (13) | 30 (13) | 28 (12)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Arterial Pressure
Description: Mean arterial blood pressure was calculated from non-invasive systolic and diastolic arm measurements.
Time Frame: Baseline and 28 days
Population: Mean arterial blood pressure values were not available at all time points for every patient. Data on subjects who completed the study is presented here and may not reflect changes seen in a larger population.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Change From Base 1 to PVC Suppression: This arm will undergo attempted PVC suppression using flecainide for 28 days and then undergo no PVC suppression using placebo for 28 days.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  Change in BP values from baseline to PVC suppression in the group that received flecainide (PVC suppression) first.
- Change From Base 2 to no PVC Suppression: This arm will undergo attempted PVC suppression using flecainide for 28 days and then undergo no PVC suppression using placebo for 28 days.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  Change in BP values from 2nd baseline (washout) to PVC suppression in the group that received flecainide (PVC suppression) first.
- Change From Base 1 to no PVC Suppression: This arm will undergo no PVC suppression using placebo for 28 days and then undergo attempted PVC suppression using flecainide for 28 days.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  Change in BP values from first baseline to no PVC suppression in the group that received placebo (no PVC suppression) first.
- Change From Base 2 to PVC Suppression: This arm will undergo no PVC suppression using placebo for 28 days and then undergo attempted PVC suppression using flecainide for 28 days.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  Change in BP values from 2nd baseline (washout) to PVC suppression in the group that received placebo (no PVC suppression) first.
Arm/Group | Change From Base 1 to PVC Suppression | Change From Base 2 to no PVC Suppression | Change From Base 1 to no PVC Suppression | Change From Base 2 to PVC Suppression
Number analyzed (Participants) | 3 | 3 | 4 | 4
mmHg | 2 (2) | 1 (4) | 3 (11) | -4 (8)

2. Secondary Outcome: Change in Muscle Sympathetic Nerve Activity
Description: Muscle sympathetic nerve activity was measured as number of bursts of neural activity per 100 heart beats.
Time Frame: Baseline and 28 days
Population: SNA values were not obtained in many of the participants in various groups above due to technical difficulties. Data on subjects who underwent the measurement are presented here and may not reflect changes seen in a larger population.
Measure: Number; unit: bursts / 100 heartbeats
Groups:
- Change From Base 1 to PVC Suppression: This arm will undergo attempted PVC suppression using flecainide for 28 days and then undergo no PVC suppression using placebo for 28 days.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  Change in SNA values from baseline to PVC suppression in the group that received flecainide (PVC suppression) first.
- Change From Base 2 to no PVC Suppression: This arm will undergo attempted PVC suppression using flecainide for 28 days and then undergo no PVC suppression using placebo for 28 days.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  Change in SNA values from 2nd baseline (washout) to PVC suppression in the group that received flecainide (PVC suppression) first.
- Change From Base 1 to no PVC Suppression: This arm will undergo no PVC suppression using placebo for 28 days and then undergo attempted PVC suppression using flecainide for 28 days.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  Change in SNA values from first baseline to no PVC suppression in the group that received placebo (no PVC suppression) first.
- Change From Base 2 to PVC Suppression: This arm will undergo no PVC suppression using placebo for 28 days and then undergo attempted PVC suppression using flecainide for 28 days.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  Change in SNA values from 2nd baseline (washout) to PVC suppression in the group that received placebo (no PVC suppression) first.
Arm/Group | Change From Base 1 to PVC Suppression | Change From Base 2 to no PVC Suppression | Change From Base 1 to no PVC Suppression | Change From Base 2 to PVC Suppression
Number analyzed (Participants) | 1 | 1 | 1 | 1
bursts / 100 heartbeats | 1 | -10 | -3 | 15

3. Other Pre Specified Outcome: Change in Baroreflex Gain
Description: Arterial baroreflex gain is calculated as slope of the relationship between cardiac cycle length and the corresponding change in systolic blood pressure.
Time Frame: Baseline and 28 days
Population: Arterial baroreflex gain values were not available at all time points. In one subject, gain could not be calculated because they were in bigeminy. Data on subjects who completed the study is presented here and may not reflect changes seen in a larger population.
Measure: Mean (Standard Deviation); unit: ms/mmHg
Groups:
- Change From Base 1 to PVC Suppression: This arm will undergo attempted PVC suppression using flecainide for 28 days and then undergo no PVC suppression using placebo for 28 days.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  Change in baroreflex gain values from baseline to PVC suppression in the group that received flecainide (PVC suppression) first.
- Change From Base 2 to no PVC Suppression: This arm will undergo attempted PVC suppression using flecainide for 28 days and then undergo no PVC suppression using placebo for 28 days.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  Change in baroreflex gain values from 2nd baseline (washout) to PVC suppression in the group that received flecainide (PVC suppression) first.
- Change From Base 1 to no PVC Suppression: This arm will undergo no PVC suppression using placebo for 28 days and then undergo attempted PVC suppression using flecainide for 28 days.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  Change in baroreflex gain values from first baseline to no PVC suppression in the group that received placebo (no PVC suppression) first.
- Change From Base 2 to PVC Suppression: This arm will undergo no PVC suppression using placebo for 28 days and then undergo attempted PVC suppression using flecainide for 28 days.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  Change in baroreflex gain values from 2nd baseline (washout) to PVC suppression in the group that received placebo (no PVC suppression) first.
Arm/Group | Change From Base 1 to PVC Suppression | Change From Base 2 to no PVC Suppression | Change From Base 1 to no PVC Suppression | Change From Base 2 to PVC Suppression
Number analyzed (Participants) | 3 | 3 | 4 | 4
ms/mmHg | 4 (1) | 6 (2) | 8 (5) | 15 (7)

ADVERSE EVENTS:
Groups:
- Base 1 to PVC Suppression: This arm will undergo attempted PVC suppression using flecainide for 28 days and then undergo no PVC suppression using placebo for 28 days.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  Adverse events during baseline to PVC suppression in the group that received flecainide (PVC suppression) first.
- Base 2 to no PVC Suppression: This arm will undergo attempted PVC suppression using flecainide for 28 days and then undergo no PVC suppression using placebo for 28 days.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  Adverse events during 2nd baseline (washout) to PVC suppression in the group that received flecainide (PVC suppression) first.
- Base 1 to no PVC Suppression: This arm will undergo no PVC suppression using placebo for 28 days and then undergo attempted PVC suppression using flecainide for 28 days.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  Adverse events during first baseline to no PVC suppression in the group that received placebo (no PVC suppression) first.
- Base 2 to PVC Suppression: This arm will undergo no PVC suppression using placebo for 28 days and then undergo attempted PVC suppression using flecainide for 28 days.
  No PVC Suppression using Placebo: Placebo (sugar pills) will be given to result in no alteration in PVC burden.
  PVC Suppression using Flecainide: Flecainide will be administered to result in a reduction in PVC burden.
  Adverse events during 2nd baseline (washout) to PVC suppression in the group that received placebo (no PVC suppression) first.
Arm/Group | Base 1 to PVC Suppression | Base 2 to no PVC Suppression | Base 1 to no PVC Suppression | Base 2 to PVC Suppression
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/4

LIMITATIONS AND CAVEATS:
This study was terminated prematurely due to a loss of staff available to make the technical measurements involved. The small number of data points available lead us to conclude the data is uninterpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes